CLINICAL TRIAL: NCT04827004
Title: A Open-label, Single-center, Single-arm Phase II Study of Anlotinib Hydrochloride Capsules in Subjects With Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Anlotinib Hydrochloride Capsules in Subjects With Diffuse Large B-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-20-II
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-07

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride Capsules (Experimental): This is a multi-target receptor tyrosine kinase inhibitor.
  Interventions: Drug: Anlotinib Hydrochloride Capsules

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsules — Anlotinib capsules given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).

SUMMARY:
This is an open-label, single-center, single-arm study to evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules in subjects with diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years old; Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, life expectancy≥ 12 weeks.

  2. Histopathologically confirmed diffuse large B-cell lymphoma (DLBCL) . 3. Has received at least 2 lines of systemic treatment. 4. At least one measurable lesion in vertical directions(based on Lugano 2014). 5.Adequate organ system function. 6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ; No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

  7. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. DLBCL transformed from indolent lymphoma (such as FL), primary testicular DLBCL, primary central nervous system lymphoma, mixed lymphoma (such as B cell lymphoma that cannot be classified between HL and DLBCL) Tumor, etc.), Richter's transformed DLBCL.

  2. Has central nervous system (CNS) invasion. 3. Has received vascular endothelial growth inhibitor, such as sunitinib, sorafenib, pazopanib, imatinib, famitinib, apatinib, anlotinib and so on.

  4. Has other malignancies (except cured skin basal cell carcinoma and cervical carcinoma in situ) within 3 years.

  5. Has a history of immunodeficiency. 6. Has multiple factors affecting oral medication. 7.Has uncontrollable or important cardiovascular disease. 8.Has any severe and/or uncontrolled diseases. 9. Has received surgery, or unhealed wounds within 4 weeks before the first administration.

  10. Has received systemic steroid therapy within 7 days before the first administration.

  11. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear.

  12. Has any bleeding symptoms or treated with anticoagulants or vitamin K antagonists.

  13. Has arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident including transient ischemic attack, deep vein thrombosis and pulmonary embolism.

  14. Has psychotropic substances abuse or a mental disorder. 15. Has received autologous hematopoietic stem cell transplantation within 3 months before the first administration, or have received allogeneic hematopoietic stem cell transplantation, or have graft-versus-host reaction.

  16. Has received other anti-tumor therapy within 4 weeks before the first administration.

  17.According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

  18. Unsuitable for anlotinib hydrochloride.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 48 weeks
  PFS defined as the time from first medication until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 48 weeks
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Duration of Response (DOR) | up to 48 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China